CLINICAL TRIAL: NCT00135863
Title: Intraperitoneal Low Molecular Weight Heparin in Peritoneal Dialysis
Brief Title: MesoHep II: Intraperitoneal Low Molecular Weight Heparin in Peritoneal Dialysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Ribe County Hospital (Other)
Collaborators: LEO Pharma (Industry); Coloplast A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MesoHep II; 2564-03; 2612-2459
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2004-01

CONDITIONS: Inflammation; Nutrition; Peritoneal Dialysis
MeSH Terms: conditions — Inflammation | interventions — Tinzaparin

INTERVENTIONS:
Drug: tinzaparin

SUMMARY:
Patients with end stage renal disease (ESRD) who use peritoneal dialyses with Physioneal(R) (Baxter A/S, Denmark) were allocated to inject either placebo or tinzaparin daily into the morning dialysis bag. Active medication, as well as placebo, was added for three months separated by a one month washout period. At the beginning and end of each treatment period peritoneal equilibrations tests (PE-tests), Kt/V, blood and dialysate samples were analyzed. We, the researchers at Ribe County Hospital, set out to examine inflammation (local and systemic), nutrition and ultrafiltration.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease
* Peritoneal dialysis without complication for minimum of three months
* 18 years or above
* Informed consent

Exclusion Criteria:

* Known coagulatory defects including anticoagulation therapy
* Known bleeding tendency
* Peritonitis within two months prior to inclusion
* Pregnancy
* Breast feeding
* Active infection
* Non-informed consent
* Allergy to heparin or prior heparin induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2004-05; Study Completion 2005-05

PRIMARY OUTCOMES:
Grade of inflammation, local and systemic

SECONDARY OUTCOMES:
Vascular compliance
Nutritional state
Efficacy of Peritoneal Dialysis
Change in local cellular distribution
Change in local and systemic generation of thrombi

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Petersen, MD, Study Chair — Ribe County Hospital, Department of Nephrology; Mikkel B Rasmussen, MD, Principal Investigator — Ribe County Hospital, Department of Nephrology
Locations (1):
- Ribe County Hospital, Esbjerg, Ribe, Denmark